CLINICAL TRIAL: NCT03116724
Title: Direct Measurement of Ideal Depth of Central Line for Right Internal Jugular Venous Catheterization in Adults
Brief Title: Direct Measurement of Ideal Depth of Central Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Jiwon Lee, assistant professor, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ideal depth of central line
Record Dates: First submitted 2017-04-04; First posted 2017-04-17 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Patient Safety During Central Venous Catheterization
Keywords: catheterization, central venous; jugular veins; echocardiography, transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVC catheterization through Rt. IJV (Experimental): The depth of central venous catheter during central venous catheterization through Rt. IJV will be decided by using real-time TEE.
  The position of tip of CVC will be guided by TEE to fit the tip at 2 cm away from the junction between right atrium and superior vena cava.
  Interventions: Procedure: central venous catheterization through Rt. IJV

INTERVENTIONS:
Procedure: central venous catheterization through Rt. IJV — * insertion at the intersection of the cricoid cartilage level and the triangular point where the sternal head of the SCM muscle meets the clavicular head
  * placement of the tip of the catheter 2 cm away from the junction between right atrium and superior vena cava using TEE
  * measurement of the depth of the catheter at insertion point

SUMMARY:
Total of 89 patients undergoing elective cardiac surgery will be enrolled.

Right CVC insertion begins at their intersection of the cricoid cartilage level and the triangular point where the sternal head of the SCM muscle meets the clavicular head. After insertion the central venous catheter through the right internal jugular vein and positioning it, the location of the tip of the central venous catheter will be confirmed by TEE.

DETAILED DESCRIPTION:
Investigator confirms the location of the 2 cm from the junction between right atrium and superior vena cava to the end of the tip of the catheter using TEE, and measures the insertion depth of the catheter at insertion point. It is possible to find the ideal central venous catheter insertion depth in actual clinical practice in adult patient.

The ideal central venous catheter insertion depth can be measured accurately when the end of the central venous catheter is monitored with transesophageal ultrasonography, and it can be derived a meaningful formula for predicting the ideal central venous insertion depth from the patient's height .

ELIGIBILITY:
Inclusion Criteria:

* adult patient over 18 years of age undergoing cardiac surgery under general anesthesia, requiring central venous catheter insertion through the right internal jugular vein and insertion of a TEE probe

Exclusion Criteria:

* Patients who disagree with the study.
* Patients who had difficulty in inserting the central line through the right internal jugular vein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
depth of the central venous catheter in right internal jugular vein | at time of insertion of the central venous catheter

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Lee, Dr., Principal Investigator — Dongsan Medical Center
Locations (1):
- Dongsan medical center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No